CLINICAL TRIAL: NCT06973499
Title: Exploratory Study of the Microbiome of Upper Gastrointestinal in the Pathogenesis of Multiple Primary Lung Cancer
Status: Completed | Type: Observational
Sponsor: Beijing Haidian Hospital (Other)
Responsible Party: Principal Investigator, Huang Yuqing, Director, Beijing Haidian Hospital
Other Study IDs: BHHMEC-XM-2022-42
Record Dates: First submitted 2022-06-25; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Multiple Primary Lung Cancer; Microbial Colonization
Keywords: Multiple Primary Lung Cancer; Microbiome
MeSH Terms: conditions — Communicable Diseases | interventions — Symptom Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples were collected aseptically from seven anatomical sites:
  Upper respiratory tract: Nasal swabs (inserted to the nasopharynx, rotated 3×, stored in RNase-free tubes at -70°C).
  Oral cavity: Pharyngeal swabs (8-10 s swabbing, liquid nitrogen snap-freezing).
  Lower respiratory tract: Bronchoalveolar lavage fluid (BALF, ≥1 mL) and protected specimen brush samples via bronchoscopy.
  Upper gastrointestinal (UGI) tract: Gastric fluid (≥1 mL) via gastroscopy.
  Lung nodules and adjacent tissues: Fresh surgical specimens (≥150 mg) rinsed with PBS, flash-frozen in liquid nitrogen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study arm: 1. Microbial samples of oral cavity, upper and lower respiratory tract, upper digestive tract, lung lavage fluid, malignant pulmonary nodules and their adjacent sites, pathological samples and blood samples of patients with multiple primary lung cancer should be collected.
  2. Blood samples were tested for T and B lymphocyte subsets, NK cell percentage and immune factors. Metagenomic sequencing (16S rDNA sequencing at malignant pulmonary nodules) was performed on the bacterial community samples from different parts, and exome and transcriptome sequencing were performed on the lesion and its adjacent tissues to obtain the genome mutation and transcriptome information of the corresponding samples.
  3. In view of the above key characteristics, differentially expressed genes, pathway analysis and functional module construction were carried out to screen biologically important modules and genes related to lung cancer mutation and bacterial community microenvironment.
  Interventions: Diagnostic Test: Microbiome Profiling and Symptom Assessment

INTERVENTIONS:
Diagnostic Test: Microbiome Profiling and Symptom Assessment — GERD symptom assessment: Standardized GERD-Q questionnaire to evaluate reflux symptoms (heartburn, acid regurgitation) and high-risk behaviors.
  Microbiome analysis: 16S rDNA sequencing of upper gastrointestinal and intratumoral microbiota.

SUMMARY:
This is an exploratory, single-center, being conducted at Beijing Haidian Hospital in order to detect the relationship between microbiome of upper gastrointestinal and pathogenesis of multiple primary lung cancer.

DETAILED DESCRIPTION:
This study intends to analyze the bacterial community structure of respiratory tract, upper digestive tract, lesion and adjacent to cancer in patients with multiple primary lung cancer, and to explore the association between upper digestive tract bacterial community and lung microecology, in order to find the characteristics of upper digestive tract bacterial strains involved in regulating lung cancer microenvironment, and explore the possible interaction mechanism between upper digestive tract bacterial community and lung cancer gene mutation.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age (including 18 years of age, male or female) and voluntarily signed informed consent;
2. Chest CT imaging showed at least 2 pulmonary nodules with a diameter of less than 3cm in ipsilateral lung, and imaging diagnosis of highly suspicious multiple primary lung cancer
3. No surgical contraindication, surgical resection is feasible, and postoperative pathology is diagnosed as multiple primary lung cancer according to Martini and Melamed criteria and gene testing
4. The amount of at least 2 or more tissues removed from multiple pulmonary nodules must meet the requirements of pathological diagnosis, molecular detection and microflora detection

Exclusion Criteria:

1. under 18 years of age (excluding 18 years of age, male or female) or unwilling to sign informed consent;
2. severe heart, liver, brain, kidney and other important organ diseases and bone marrow hematopoietic dysfunction;
3. Preoperative examination of patients who cannot tolerate surgical resection
4. Patients who received antibiotics within 1 week before surgery E) Resected multiple pulmonary nodules with pathologically proven lung cancer of less than 2 patients
5. Multiple nodules resected were confirmed to be metastases, not primary lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Multiple primary lung cancer patients
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Microbial homology between upper gastrointestinal (UGI) microbiota and intratumoral microbiota | Sequencing and analysis will be completed within 6 months after sample collection.
  Based on 16S rDNA sequencing data, calculate the Bray-Curtis similarity index between the intratumoral microbiota and the patient's own upper gastrointestinal (UGI) microbiota. Use SourceTracker2 to quantify the contribution of UGI microbiota to the intratumoral microbiota. Apply PERMANOVA analysis to compare the differences in microbiota similarity between the MPLC and SPLC groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yuqing Huang, M.D., Study Director — Beijing Haidian Hospital
Locations (1):
- Beijing Haidian Hospital, Beijing, China, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peters BA, Hayes RB, Goparaju C, Reid C, Pass HI, Ahn J. The Microbiome in Lung Cancer Tissue and Recurrence-Free Survival. Cancer Epidemiol Biomarkers Prev. 2019 Apr;28(4):731-740. doi: 10.1158/1055-9965.EPI-18-0966. Epub 2019 Feb 7. PMID 30733306